CLINICAL TRIAL: NCT05706064
Title: Survey of COVID-19 Infection
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, LingTao, Professor in Cardiology, Director of the department of Cardiology, Xijing Hospital
Other Study IDs: Survey of COVID-19 infection
Record Dates: First submitted 2023-01-29; First posted 2023-01-31 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: COVID-19; Infections
MeSH Terms: conditions — COVID-19; Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 Infection

SUMMARY:
Using online questionnaires, we will obtain data regarding COVID-19 infection and treatment, including incidence rate, hospitalization rate, severity of the infection, medications, mortality rate, etc, in both hospital and communities after the change of disease control policy in China.

ELIGIBILITY:
Inclusion Criteria:

* N/A

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All population from hospital and community
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 6 months
  Quickly obtain the all-cause mortality in patients with COVID-19

SECONDARY OUTCOMES:
Incidence rate of COVID-19 infection | 6 months
  Incidence rate of COVID-19 infection
Medication for COVID-19 treatment | 6 months
  Any medication for COVID-19 treatment
Hospitalization rate due to COVID-19 infection | 6 months
  Hospitalization rate due to COVID-19 infection
Severity of COVID-19 infection | 6 months
  severity of the COVID-19 infection

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, MD, Ph.D., Study Chair — Xijing Hospital; Chao Gao, MD, Ph.D., Study Chair — Xijing Hospital
Locations (1):
- Ling Tao, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No